CLINICAL TRIAL: NCT03730662
Title: Efficacy and Safety of LY3298176 Once Weekly Versus Insulin Glargine in Patients With Type 2 Diabetes and Increased Cardiovascular Risk (SURPASS-4)
Brief Title: A Study of Tirzepatide (LY3298176) Once a Week Versus Insulin Glargine Once a Day in Participants With Type 2 Diabetes and Increased Cardiovascular Risk
Acronym: SURPASS-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17072; I8F-MC-GPGM (Other: Eli Lilly and Company); 2018-002618-11 (EudraCT Number)
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GIP; GLP-1; glucose metabolism disorders; metabolic diseases; endocrine system diseases; cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — Tirzepatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg Tirzepatide (Experimental): 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): 10 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): 15 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- Insulin Glargine (Active Comparator): Insulin glargine administered SC once a day. Doses were individualized and titrated according to protocol-defined targets.
  The starting dose of insulin glargine was 10 IU/day at bedtime, titrated to a FBG <100 mg/dL, following a treat-to-target (TTT) algorithm.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Tirzepatide — Administered SC.
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Insulin Glargine — Administered SC
  Arms: Insulin Glargine

SUMMARY:
The purpose of the trial is to assess the efficacy and safety of tirzepatide taken once a week to insulin glargine taken once daily in participants with type 2 diabetes and increased cardiovascular risk. The study will last about 108 weeks and may include up to 30 visits.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Have been diagnosed with type 2 diabetes mellitus (T2DM)
* Have HbA1c between ≥7.5% and ≤10.5%
* Be on stable treatment with unchanged dose of at least 1 and no more than 3 types of oral antihyperglycemic drugs, which may only include metformin, SGLT-2 inhibitors, and/or sulfonylureas for at least 3 months before screening
* Have increased risk for cardiovascular (CV) events
* Be of stable weight (± 5%)
* Have a BMI ≥25 kilograms per meter squared (kg/m2) at screening

Exclusion Criteria

Participants must not:

* Have type 1 diabetes mellitus
* Have had chronic or acute pancreatitis any time prior to study entry
* Have proliferative diabetic retinopathy or diabetic maculopathy or nonproliferative diabetic retinopathy requiring immediate or urgent treatment
* Have disorders associated with slowed emptying of the stomach, or have had any stomach surgeries for the purpose of weight loss
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or blood alanine transaminase (ALT) enzyme level >3.0 times the upper limit of normal (ULN) for the reference range, as determined by the central laboratory. Participants with nonalcoholic fatty liver disease (NAFLD) are eligible for participation in this trial only if there ALT level is ≤3.0 the ULN for the reference range
* Have had a heart attack, stroke, or hospitalization for congestive heart failure in the past 2 months
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2
* Have been taking any other diabetes medicines other than metformin, SGLT-2 inhibitors, and/or sulfonylureas during the last 3 months
* Have been taking weight loss drugs, including over-the-counter medications during the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2002 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (215):
- United States (73):
  - Advanced Research Center, Anaheim, California
  - Valley Clinical Trials, Inc., Covina, California
  - Marin Endocrine Associates, Greenbrae, California
  - National Research Institute, Huntington Park, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - First Valley Medical Group, Lancaster, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Monterey Endocrine & Diabetes Institute, Inc., Monterey, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Medical Group Inc, Palm Springs, California
  - Havana Research Institute, Pasadena, California
  - Western University of Health Sciences, Pomona, California
  - LCGK Research, San Carlos, California
  - Olive View Medical Center, Sylmar, California
  - University Clinical Investigators, Inc., Tustin, California
  - Touro University, Vallejo, California
  - Coastal Metabolic Research Centre, Ventura, California
  - Diablo Clinical Research, Walnut Creek, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - ALL Medical Research, LLC, Cooper City, Florida
  - Advanced Pharma Research, Cutler Bay, Florida
  - South Florida Wellness & Clinical Research Institute, Margate, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Primary Care Specialists, LLC, Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Saltzer Medical Group. P.A., Nampa, Idaho
  - Northwestern Feinberg School of Medicine, Chicago, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois
  - University of Iowa Hospital & Clinic, Iowa City, Iowa
  - Iowa Diabetes Research, West Des Moines, Iowa
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - Robley Rex VAMC, Louisville, Kentucky
  - NECCR PrimaCare Research, LLC, Fall River, Massachusetts
  - AA Medical Research Center, Flint, Michigan
  - Troy Internal Medicine, PC, Troy, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Montana Medical Research, Inc, Missoula, Montana
  - Palm Research Center, Las Vegas, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - PharmQuest, Greensboro, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Ohio State Univ College Of Medicine, Columbus, Ohio
  - Aventiv Research, Columbus, Ohio
  - Intend Research, Norman, Oklahoma
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Capital Area Research, Camp Hill, Pennsylvania
  - Detweiler Family Medicine, Lansdale, Pennsylvania
  - Capital Area Research, Newport, Pennsylvania
  - Parkside Family Medical, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians- Bower Hill, Pittsburgh, Pennsylvania
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - The Research Center of the Upstate, Mauldin, South Carolina
  - Holston Medical Group Clinical Research, Kingsport, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - PCP for Life, Houston, Texas
  - BFHC Research, San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Alpine Research Organization, Farmington, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Private: Dr. Larry Stonesifer, Federal Way, Washington
  - Capital Clinical Research Center, Olympia, Washington
  - Walla Walla Clinic, Walla Walla, Washington
- Argentina (15):
  - Centro de Investigaciones Metabólicas (CINME), CABA, Buenos Aires
  - Mautalen Salud e Investigación - Servicio de Endocrinología, CABA, Buenos Aires
  - Investigaciones Medicas IMOBA S.R.L., Caba, Buenos Aires
  - CEDIC-Centro de Investigaciones Clinicas, Caba, Buenos Aires
  - CEMEDIC, CABA, Buenos Aires
  - Centro Medico Dr Laura Maffei Investigacion Clinica Aplicada, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Centro de Investigacion y Prevencion Cardiovascular (CIPREC), Ciudad Autonoma de, Buenos Aires
  - CIPADI, Godoy Cruz, Mendoza Province
  - AXISMED SRL - Bioclinica Research Network, Buenos Aires
  - Centro Médico Viamonte, Ciudad Autonoma de Buenos Aire
  - Instituto Centenario, Ciudad Autonoma de Buenos Aire
  - Cemediab - Centro Médico Diabetológico Dr. Alejandro Chertkoff, Ciudad Autonoma de Buenos Aire
  - Centro Diabetologico Dr Waitman, Córdoba
  - Centro Medico Privado San Vicente Diabetes, Córdoba
  - Cent Priva Especiali Médicas Ambulatorias Inve Clin CEMAIC, Córdoba
- Australia (15):
  - Paratus Clinical Blacktown Clinic, Blacktown, New South Wales
  - Campbelltown Medical & Dental Centre, Campbelltown, New South Wales
  - Paratus Clinical Kanwal Clinic, Kanwal, New South Wales
  - The AIM Centre, Merewether, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - CORE Research Group Pty Ltd, Brisbane, Queensland
  - Morayfield Medical and Dental Centre, Morayfield, Queensland
  - AusTrials Pty Ltd, Sherwood, Queensland
  - Victoria Point Medical and Dental Centre, Victoria Point, Queensland
  - GP Plus Marion, Oaklands Park, South Australia
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Forest Hill Medical and Dental Centre, Forest Hill, Victoria
  - Barwon Health - The Geelong Hospital, Geelong, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Brazil (9):
  - Instituto de Ensino e Pesquisa Clinica do Ceara, Fortaleza, Ceará
  - Cedoes Centro Diagnostico Pequisa Osteoporose E Santo Ltd, Vitória, Espírito Santo
  - Centro de Pesquisa Clinica do Brasil, Brasília, Federal District
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - CCBR Brasil Centro de Analises e Pesquisas Clínicas LTDA, Rio de Janeiro, Rio de Janeiro
  - CPQuali Pesquisa Clínica Ltda., São Paulo, São Paulo
  - Cpclin Centro de Pesquisas Clinicas, São Paulo, São Paulo
  - Centro de Pesq. em Diabetes e Doencas Endocrino Metabol., Fortaleza
  - Dr. Consulta Clínica Médica LTDA, São Paulo
- Canada (19):
  - LMC Manna Research, Calgary, Alberta
  - C-Health Diabetes and Endocrinology Clinic Calgary, Calgary, Alberta
  - Synergy Medical Research, Sherwood Park, Alberta
  - LMC Endocrinology Centres Ltd., Barrie, Ontario
  - LMC Endocrinology Centers Brampton, Brampton, Ontario
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - LMC Endocrinology Centres Ltd., Concord, Ontario
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Milestone Research Inc., London, Ontario
  - LMC Endocrinology Centres Ltd., Nepean, Ontario
  - Bluewater Clinical Research Group Inc, Sarnia, Ontario
  - Canadian Centre for Research on Diabetes, Smiths Falls, Ontario
  - Manna Research, Inc., Stoney Creek, Ontario
  - LMC Endocrinology Centres Ltd., Toronto, Ontario
  - Sameh Fikry Medicine Professional Corporation, Waterloo, Ontario
  - Q & T Research Outaouais, Gatineau, Quebec
  - Centre De Recherche Clinique De Laval, Laval, Quebec
  - Manna Research (Quebec), Lévis, Quebec
  - LMC Endocrinology Centres Ltd., Saint-Laurent, Quebec
- Greece (5):
  - Iatriko Palaiou Falirou, Medical Center, Palaió Fáliro, Athens
  - Thermi Clinic, Thermi, Thessaloniki
  - University General Hospital of Larissa, Larissa
  - AHEPA Hospital, Thessaloniki
  - Euromedica - General Clinic of Thessaloniki, Thessaloniki
- Israel (9):
  - Ha'Emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sakhnin Community Clinic, Clalit Health Services, Sakhnin
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Mexico (6):
  - Instituto Jalisciense de Investigacion en Diabetes y Obesida, Guadalajara, Jalisco
  - Diseno y Planeacion en Investigacion Medica S.C., Guadalajara, Jalisco
  - Unidad Medica para la Salud Integral (UMSI), Monterrey, Nuevo León
  - St. Lucas Clinical Research Center, Merida, State of Mexico
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasc, Tampico, Tamaulipas
  - Investigacion en Salud y Metabolismo S.C, Chihuahua City
- Poland (11):
  - Centralny Szpital Kliniczny MSWiA Klinika Dermatologiczna, Warsaw, Masovian Voivodeship
  - Poradnia Diabetologiczna SN ZOZ Lege Artis, Bialystok
  - NZOZ Diab-Endo-Met, Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - NZOZ CenterMed Lublin, Lublin
  - Gabinety Terpa, Lublin
  - NZOZ Przychodnia Specjalistyczna MEDICA, Lublin
  - Praktyka Lekarska, Poznan
  - Nzoz Neuro - Kard, Poznan
  - NZOZ Przychodnia Specjalistyczna Henryk RudzkiAndrzej Wittek, Ruda Śląska
  - Woj. Zesp. Spec. Opieki Zdrowotnej, Wroclaw
- Puerto Rico (7):
  - Manati Center for Clinical Research Inc, Manatí, PR
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - Research and Cardiovascular Corp., Ponce, PR
  - University Of Puerto Rico, Rio Pedras, PR
  - GCM Medical Group PSC, San Juan, PR
  - Consultorio Medico, San Juan, PR
  - Emanuelli Research & Development Center, LLC, Arecibo
- Romania (9):
  - SC Gama Diamed SRL, Mangalia, Constanța County
  - Spitalul Judetean de Urgenta Satu Mare, Satu Mare, Jud Satu-Mare
  - CMI DNBM Dr. Pop Lavinia, Baia Mare, Maramureş
  - Cosamext SRL, Târgu Mureş, Mureș County
  - Centrul Medical Dr. Negrisanu, Timișoara, Timiș County
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed SRL, Brasov
  - Cabinetul Medical Nicodiab SRL, Bucharest
  - SC Nutrilife SRL, Bucharest
  - Milena Sante SRL, Galati
- Russia (10):
  - Regional Clinical Hospital, Saratov, Russian Federation
  - Arkhangelsk the first city clinical hospital, Arkhangelsk
  - FSBI Endocrinological Research Center of the MOH of the ROF, Moscow
  - Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Ryazan Regional Clinincal Cardiology Dispensary, Ryazan
  - City Hospital of Saint Martyr Elizabeth, Saint Petersburg
  - Medical Military Academy, Saint Petersburg
  - City Consultative and Diagnostic Center, Saint Petersburg
  - SPb GUZ "Diagnostic Center #85", Saint Petersburg
  - Research & Practice Ltd, Yaroslavl
- Slovakia (6):
  - Human care s.r.o., Košice, Slovak Republic
  - MediVet s.r.o., Malacky, Slovak Republic
  - Areteus s.r.o., Trebišov, Slovak Republic
  - DIA-MED CENTRUM s.r.o., Púchov
  - Tatratrial s.r.o., Rožňava
  - MEDI-DIA s.r.o., Sabinov
- Spain (12):
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital de la Ribera, Alzira, Valencia
  - Complexo Hospitalario Universitario A Coruña, CHUAC, A Coruña
  - Instituto de Ciencias medicas, Alicante
  - Centro Periférico de Especialidades Bola Azul, Almería
  - Hospital Quironsalud Barcelona- END, Barcelona
  - Hospital Clinico Universitario San Cecilio, Granada
  - Centro Especialidades San Jose Obrero (Barbarela), Málaga
  - Clinica Juaneda, Palma de Mallorca
  - Clinica Nuevas Tecnologias en Diabetes y Endocrinologia, Seville
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (9):
  - Cardinal Tien Hospital, Sindian City, Taipei
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Kuang Tien General Hospital, Taichung County
  - National Cheng Kung University Hospital, Tainan
  - Chi-Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] De Block C, Peleshok J, Wilding JPH, Kwan AYM, Rasouli N, Maldonado JM, Wysham C, Liu M, Aleppo G, Benneyworth BD. Post Hoc Analysis of SURPASS-1 to -5: Efficacy and Safety of Tirzepatide in Adults with Type 2 Diabetes are Independent of Baseline Characteristics. Diabetes Ther. 2025 Jan;16(1):43-71. doi: 10.1007/s13300-024-01660-0. Epub 2024 Nov 12. PMID 39531161
- [Derived] Boye KS, Sapin H, Dong W, Williamson S, Lee CJ, Thieu VT. Improved Glycaemic and Weight Management Are Associated with Better Quality of Life in People with Type 2 Diabetes Treated with Tirzepatide. Diabetes Ther. 2023 Nov;14(11):1867-1887. doi: 10.1007/s13300-023-01457-7. Epub 2023 Sep 5. PMID 37668888
- [Derived] Boye KS, Thieu VT, Sapin H, Lee CJ, Lando LF, Brown K, Bray R, Wiese RJ, Patel H, Rodriguez A, Yu M. Patient-Reported Outcomes in People with Type 2 Diabetes Receiving Tirzepatide in the SURPASS Clinical Trial Programme. Diabetes Ther. 2023 Nov;14(11):1833-1852. doi: 10.1007/s13300-023-01451-z. Epub 2023 Aug 1. PMID 37526908
- [Derived] Heerspink HJL, Sattar N, Pavo I, Haupt A, Duffin KL, Yang Z, Wiese RJ, Tuttle KR, Cherney DZI. Effects of tirzepatide versus insulin glargine on kidney outcomes in type 2 diabetes in the SURPASS-4 trial: post-hoc analysis of an open-label, randomised, phase 3 trial. Lancet Diabetes Endocrinol. 2022 Nov;10(11):774-785. doi: 10.1016/S2213-8587(22)00243-1. Epub 2022 Sep 21. PMID 36152639
- [Derived] Sattar N, McGuire DK, Pavo I, Weerakkody GJ, Nishiyama H, Wiese RJ, Zoungas S. Tirzepatide cardiovascular event risk assessment: a pre-specified meta-analysis. Nat Med. 2022 Mar;28(3):591-598. doi: 10.1038/s41591-022-01707-4. Epub 2022 Feb 24. PMID 35210595
- [Derived] Del Prato S, Kahn SE, Pavo I, Weerakkody GJ, Yang Z, Doupis J, Aizenberg D, Wynne AG, Riesmeyer JS, Heine RJ, Wiese RJ; SURPASS-4 Investigators. Tirzepatide versus insulin glargine in type 2 diabetes and increased cardiovascular risk (SURPASS-4): a randomised, open-label, parallel-group, multicentre, phase 3 trial. Lancet. 2021 Nov 13;398(10313):1811-1824. doi: 10.1016/S0140-6736(21)02188-7. Epub 2021 Oct 18. PMID 34672967
- See also: A Study of Tirzepatide (LY3298176) Once a Week Versus Insulin Glargine Once a Day in Participants With Type 2 Diabetes and Increased Cardiovascular Risk — https://trials.lillytrialguide.com/en-US/trial/740VpRcJPiyieyyWGYO2ao

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period (52 Weeks)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Started | 329 | 330 | 338 | 1005
Received at Least One Dose of Study Drug | 329 | 328 | 338 | 1000
Completed | 308 | 319 | 329 | 953
Not Completed | 21 | 11 | 9 | 52
Not completed — Adverse Event | 3 | 2 | 0 | 3
Not completed — Screen Failure | 0 | 1 | 0 | 0
Not completed — Death | 6 | 2 | 2 | 9
Not completed — Lost to Follow-up | 4 | 2 | 2 | 11
Not completed — Physician Decision | 1 | 1 | 0 | 3
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 0 | 5 | 23
Not completed — Personal Reason | 2 | 2 | 0 | 2
Period: Variable Treatment Period
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Started | 308 | 319 | 329 | 953
Completed | 294 | 312 | 313 | 882
Not Completed | 14 | 7 | 16 | 71
Not completed — Adverse Event | 1 | 2 | 0 | 7
Not completed — Death | 9 | 0 | 6 | 26
Not completed — Lost to Follow-up | 2 | 1 | 4 | 11
Not completed — Personal Reason | 0 | 2 | 1 | 6
Not completed — Physician Decision | 0 | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 4 | 17

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine | Total
Number analyzed (Participants) | 329 | 330 | 338 | 1005 | 2002
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.90 (8.56) | 63.70 (8.68) | 63.70 (8.60) | 63.80 (8.51) | 63.60 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 121 | 135 | 364 | 751
  Male | 198 | 209 | 203 | 641 | 1251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 154 | 164 | 155 | 478 | 951
  Not Hispanic or Latino | 172 | 164 | 179 | 521 | 1036
  Unknown or Not Reported | 3 | 2 | 4 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 32 | 30 | 26 | 86 | 174
  Asian | 15 | 16 | 8 | 31 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 1 | 3
  Black or African American | 13 | 18 | 11 | 34 | 76
  White | 260 | 260 | 285 | 827 | 1632
  More than one race | 8 | 6 | 5 | 24 | 43
  Unknown or Not Reported | 1 | 0 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 80 | 80 | 82 | 242 | 484
  Australia | 3 | 3 | 4 | 9 | 19
  Brazil | 42 | 41 | 42 | 125 | 250
  Canada | 8 | 9 | 7 | 27 | 51
  Greece | 7 | 5 | 7 | 19 | 38
  Israel | 4 | 5 | 5 | 15 | 29
  Mexico | 27 | 27 | 26 | 80 | 160
  Poland | 27 | 25 | 26 | 78 | 156
  Romania | 13 | 14 | 14 | 41 | 82
  Russia | 14 | 14 | 15 | 45 | 88
  Slovakia | 33 | 32 | 34 | 100 | 199
  Spain | 11 | 14 | 14 | 38 | 77
  Taiwan | 5 | 5 | 5 | 15 | 30
  United States | 55 | 56 | 57 | 171 | 339
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.52 (0.84) | 8.59 (0.91) | 8.52 (0.98) | 8.50 (0.85) | 8.52 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (10 mg and 15 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model for post-baseline measures: Variable = Baseline + Pooled Country + Baseline sodium-glucose co-transporter-2 inhibitor (SGLT-2i) use Flag (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline value, excluding participants discontinuing study drug due to inadvertent enrollment
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 289 | 291 | 887
Percentage of HbA1c | -2.43 (0.053) | -2.58 (0.053) | -1.44 (0.030)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Non-Inferiority — Although the primary objective is to establish noninferiority, sample size selection is guided by the objective of establishing superiority. The chosen sample size and randomization ratio also provides >90% power to establish superiority of 10 mg LY3298176 and 15 mg LY3298176 doses to insulin glargine in absence of confounding effects of rescue therapy for persistent severe hyperglycemia ("efficacy" estimand); p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.99, 97.5% CI 2-sided [-1.13 to -0.86]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.14, 97.5% CI 2-sided [-1.28 to -1.00]

2. Secondary Outcome: Change From Baseline in HbA1c (5 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Pooled Country + Baseline SGLT-2i use Flag (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 283 | 887
Percentage of HbA1c | -2.24 (0.053) | -1.44 (0.030)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.80, 97.5% CI 2-sided [-0.93 to -0.66]

3. Secondary Outcome: Change From Baseline in Body Weight
Description: LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline SGLT-2i use Flag (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 285 | 288 | 291 | 891
Kilograms (kg) | -7.1 (0.34) | -9.5 (0.34) | -11.7 (0.33) | 1.9 (0.19)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -9.0, 95% CI 2-sided [-9.8 to -8.3]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -11.4, 95% CI 2-sided [-12.1 to -10.6]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -13.5, 95% CI 2-sided [-14.3 to -12.8]

4. Secondary Outcome: Percentage of Participants With HbA1c of <7.0%
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Imputed data includes observed value and imputed value if endpoint measure is missing.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 326 | 321 | 334 | 978
percentage of participants | 80.98 | 88.16 | 90.72 | 50.72
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.78, 95% CI 2-sided [3.47 to 6.58]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 9.23, 95% CI 2-sided [6.31 to 13.49]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.87, 95% CI 2-sided [7.88 to 17.89]

5. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: as for outcome 3
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per Deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 281 | 283 | 288 | 880
milligram per Deciliter (mg/dL) | -50.4 (2.07) | -54.9 (2.06) | -59.3 (2.04) | -51.4 (1.17)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p = 0.672, Mixed Models Analysis; Mean Difference (Net) = 1.0, 95% CI 2-sided [-3.7 to 5.7]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p = 0.134, Mixed Models Analysis; Mean Difference (Net) = -3.6, 95% CI 2-sided [-8.2 to 1.1]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -8.0, 95% CI 2-sided [-12.6 to -3.4]

6. Secondary Outcome: Mean Change From Baseline in Daily Average 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Postmeal, Midday Premeal, Midday 2-hour Postmeal, Evening Premeal, Evening 2-hour Postmeal and Bedtime. LS mean was determined by mixed-model repeated measures (MMRM) model with variables Baseline + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline SGLT-2i use Flag (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of study drug, excluding participants discontinuing study drug due to inadvertent enrollment
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 265 | 261 | 265 | 784
mg/dL | -58.4 (1.65) | -61.1 (1.66) | -66.1 (1.66) | -46.1 (0.96)

7. Secondary Outcome: Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve From Zero to Tau (AUC 0-Tau) of Tirzepatide
Description: Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve From Zero to Tau (AUC 0-Tau) of Tirzepatide
Time Frame: 1 to 24 hours, 24 to 96 hours, or 120 to 168 hours post dose of Week 7, 15, 23, 35
Population: Pharmacokinetic samples were collected from atleast the first 150 participants at each Tirzepatide dose, all participants aged ≥70 years, and all participants with severe renal impairment or end-stage renal disease (ESRD) (estimated glomerular filtration rate [eGFR] <30 mL/min)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilitre per hour
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 326 | 324 | 334
Nanograms per millilitre per hour | 81800 (23.9) | 165000 (20.3) | 246000 (20.6)

8. Secondary Outcome: Rate of Hypoglycemia With Blood Glucose <54 Milligram/Deciliter (mg/dL) [<3.0 (Millimole/Liter (mmol/L))] or Severe Hypoglycemia
Description: The hypoglycemia events were defined by participant reported events with blood glucose <54mg/dL (<3.0 mmol/L) or severe hypoglycemia. Severe hypoglycemia is defined as an episode with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. Post-baseline comparisons between treatment and control group was evaluated using negative binomial model with variables : Number of episodes = Baseline HbA1c Group (<=8.5%, >8.5%) + Pooled Country + Baseline SGLT-2i use Flag (Yes, No) + Treatment, with log (exposure in days/365.25) as an offset variable
Time Frame: Baseline through Week 52
Population: All randomized participants who received at least one dose of study drug, excluding participants hypoglycemic events occurring after initiation of a new antihyperglycemic therapy
Measure: Mean (Standard Error); unit: Episodes/participant/365.25 days
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 329 | 328 | 338 | 1000
Episodes/participant/365.25 days | 0.10 (0.023) | 0.09 (0.025) | 0.11 (0.030) | 0.35 (0.044)

ADVERSE EVENTS:
Time Frame: Baseline Up To 2 Years
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 15/329 | 2/328 | 8/338 | 35/1000
Serious Adverse Events (participants affected / at risk) | 48/329 | 54/328 | 41/338 | 193/1000
Other Adverse Events (participants affected / at risk) | 112/329 | 158/328 | 184/338 | 192/1000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=329) | 10 mg Tirzepatide (N=328) | 15 mg Tirzepatide (N=338) | Insulin Glargine (N=1000)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 7 (7) | 3 (3) | 18 (19)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 6 (6)
Aortic valve sclerosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 5 (5) | 4 (4) | 2 (3) | 15 (16)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1/198 (1) | 0/209 (0) | 0/203 (0) | 0/636 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Necrosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Covid-19 (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 10 (10)
Covid-19 pneumonia (Infections and infestations) | 2 (2) | 6 (6) | 3 (3) | 15 (15)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hiv infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nosocomial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 10 (10)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza a virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (5) | 12 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/131 (0) | 0/119 (0) | 1/135 (1) | 0/364 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/198 (0) | 0/209 (0) | 1/203 (1) | 3/636 (3)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cranial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1) | 6 (6)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Thalamic infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/131 (0) | 0/119 (0) | 0/135 (0) | 1/364 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=329) | 10 mg Tirzepatide (N=328) | 15 mg Tirzepatide (N=338) | Insulin Glargine (N=1000)
Constipation (Gastrointestinal disorders) | 17 (17) | 14 (15) | 14 (14) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 41 (68) | 65 (128) | 74 (118) | 44 (50)
Dyspepsia (Gastrointestinal disorders) | 18 (23) | 27 (36) | 26 (36) | 13 (13)
Nausea (Gastrointestinal disorders) | 39 (104) | 53 (91) | 76 (157) | 23 (29)
Vomiting (Gastrointestinal disorders) | 16 (18) | 27 (43) | 29 (62) | 15 (16)
Covid-19 (Infections and infestations) | 13 (14) | 12 (12) | 17 (17) | 49 (49)
Nasopharyngitis (Infections and infestations) | 10 (11) | 16 (17) | 16 (19) | 65 (70)
Lipase increased (Investigations) | 10 (11) | 13 (15) | 21 (25) | 18 (18)
Decreased appetite (Metabolism and nutrition disorders) | 29 (36) | 36 (46) | 35 (43) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03730662/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03730662/SAP_001.pdf